CLINICAL TRIAL: NCT04706507
Title: Ganciclovir to Prevent Reactivation of Cytomegalovirus in Patients With Acute Respiratory Failure and Sepsis
Acronym: GRAIL^3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to increased mortality and futility analyses
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Boeckh, Professor, Vaccine and Infectious Disease Division, Fred Hutch, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RG1121219; 1UG3HL147011-01A1 (NIH); 10547 (Other: Fred Hutch)
Record Dates: First submitted 2020-12-23; First posted 2021-01-12 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Acute Respiratory Failure
MeSH Terms: interventions — Ganciclovir; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IV Ganciclovir (Experimental): 5mg/kg IV twice daily for 5 days, then followed by IV ganciclovir once daily until hospital discharge
  Interventions: Drug: IV Ganciclovir
- Placebo (Placebo Comparator): normal saline IV twice daily for 5 days, then followed by IV normal saline once daily until hospital discharge
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: IV Ganciclovir — For first 5 days, dosing of intravenous ganciclovir is 10 mg/kg daily, given as 5 mg/kg every 12 hours (adjusted for renal function). After first 5 days (up to 28 days) IV ganciclovir 5 mg/kg QD ( adjusted for renal function). A minimum interval of 6 hours is required between the first and second dose.
  Other Names: Cytovene
  Arms: IV Ganciclovir
Drug: Normal saline — For first 5 days, dosing of intravenous saline is 10 mg/kg daily, given as 5 mg/kg every 12 hours (adjusted for renal function). After first 5 days (up to 28 days) IV saline 5 mg/kg QD ( adjusted for renal function). A minimum interval of 6 hours is required between the first and second dose.
  Arms: Placebo

SUMMARY:
This is a phase 3 study designed to evaluate whether the administration of ganciclovir increases ventilator-free days in immunocompetent patients with sepsis associated acute respiratory failure. Our hypothesis is that IV ganciclovir administered early in critical illness will effectively suppress CMV reactivation in CMV seropositive adults with sepsis-associated acute respiratory failure thereby leading to improved clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* Subject/next of kin informed consent
* Age > 18 years
* CMV IgG seropositive by lateral flow assay (LFA) or standard serologic methods
* Receiving care in an ICU
* Acute respiratory failure as defined in Section 4.1.1.
* Expected to require respiratory support for at least 2 more days after randomization
* Infection confirmed or suspected by the treating clinician and felt to be the source of acute respiratory failure (Respiratory failure associated with infection confers at least 2 SOFA points above assumed baseline SOFA score of 0, thereby meeting Sepsis-3 definition).

Exclusion Criteria:

* Known or suspected immunosuppression, including:

  * HIV+ (i.e. prior positive test or clinical signs of suspicion of HIV/AIDS; a negative HIV test is not required for enrollment)
  * stem cell transplantation:

    * within 6 months after autologous transplantation or
    * within 1 years after allogeneic transplantation (regardless of immunosuppression)
    * greater than 1 year of allogeneic transplantation if still taking systemic immunosuppression or prophylactic antibiotics (e.g. for chronic graft versus host disease) Note: if details of stem cell transplantation are unknown, patients who do not take systemic immunosuppression and do not take anti-infective prophylaxis are acceptable for enrollment and randomization.
  * solid organ transplantation with receipt of systemic immunosuppression (any time)
  * cytotoxic anti-cancer chemotherapy within the past three months (Note: next-of-kin estimate is acceptable)
  * congenital immunodeficiency requiring antimicrobial prophylaxis (e.g. TMP-SMX, dapsone, antifungal drugs, intravenous immunoglobulin)
  * receipt of one or more of the following in the indicated time period (see Appendix C):

    * within 6 months: alemtuzumab, antithymocyte/antilymphocyte antibodies, or other immunosuppressive drugs associated with CMV reactivation Note: if no information on these agents is available in the history and no direct or indirect evidence exists from the history that any condition exists that requires treatment with these agents (based on the investigator's assessment), the subject may be enrolled. For all drug information, next-of-kin estimates are acceptable. See Appendix C for commonly prescribed immunosuppressive agents. Information on the use of biologics with moderate immunosuppressive effect but no known effect on CMV are permitted and will be recorded in the CRFs.
* Expected to survive < 72 hours (in the opinion of the investigator)
* Has been hospitalized for > 120 hours (subjects who are transferred from a chronic care ward, such as a rehabilitation unit, with an acute event are acceptable).
* Pregnant or breastfeeding (either currently or expected within one month). Note: for women of childbearing age (18-60 years, unless documentation of surgical sterilization [hysterectomy, tubal ligation, oophorectomy]), if a pregnancy test has not been done as part of initial ICU admission work-up, it will be ordered stat and documented to be negative before randomization. Both urine and blood tests are acceptable.
* Absolute neutrophil count < 1,000/mm3 (if no ANC value is available, the WBC must be > 2500/mm3)
* Use of anti-CMV drugs (cidofovir, letermovir, foscarnet, valganciclovir, ganciclovir) within seven (7) days of patient randomization.
* Currently enrolled in an interventional trial of an investigational therapeutic agent known or suspected to have anti-CMV activity or to be associated with significant known hematologic toxicity (prior approval required).
* At baseline patients who have both a tracheostomy, and have been on continuous 24-hour chronic mechanical ventilation.
* Patients with Child Class C Cirrhosis.
* Patients with severe (requiring home oxygen) pre-existing interstitial lung disease.
* Allergy to ganciclovir
* Incarcerated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2025-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boeckh, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (20):
- United States (20):
  - University of Colorado Denver, Denver, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Montefioure Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Wakeforest University, School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical College of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - University of Vermont College of Medicine, Burlington, Vermont
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin School of Medicine & Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 205 participants were enrolled at 19 U.S. clinical sites from June 29, 2021 until September 27, 2024 when the DSMB recommended early study closure.
Pre-assignment Details: 205 participants met the eligibility criteria. They were enrolled and randomized to study treatment simultaneously.
Groups:
- Placebo: normal saline IV twice daily for 5 days, then followed by IV normal saline once daily until hospital discharge
  IV Ganciclovir: For first 5 days, dosing of intravenous ganciclovir is 10 mg/kg daily, given as 5 mg/kg every 12 hours (adjusted for renal function). After first 5 days (up to 28 days) IV ganciclovir 5 mg/kg QD ( adjusted for renal function). A minimum interval of 6 hours is required between the first and second dose.
Period: Overall Study
Arm/Group | IV Ganciclovir | Placebo
Started | 106 | 99
Completed | 47 | 59
Not Completed | 59 | 40
Not completed — Death | 45 | 22
Not completed — Unable to adhere | 0 | 2
Not completed — Lost to Follow-up | 13 | 12
Not completed — Withdrawal of consent | 1 | 1
Not completed — Patient or LAR refuses further participation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: normal saline IV twice daily for 5 days, then followed by IV normal saline once daily until hospital discharge
  Placebo: For first 5 days, dosing of intravenous saline is 10 mg/kg daily, given as 5 mg/kg every 12 hours (adjusted for renal function). After first 5 days (up to 28 days) IV saline 5 mg/kg QD ( adjusted for renal function). A minimum interval of 6 hours is required between the first and second dose.
- Total: Total of all reporting groups
Arm/Group | IV Ganciclovir | Placebo | Total
Number analyzed (Participants) | 106 | 99 | 205
Age, Continuous [Median (Full Range); unit: years] | 63 [21 to 91] | 59 [21 to 97] | 62 [21 to 97]
Age, Customized [Count of Participants; unit: Participants]
  18 - 20 | 0 | 0 | 0
  21 - 30 | 5 | 7 | 12
  31 - 40 | 8 | 11 | 19
  41 - 50 | 13 | 14 | 27
  51 - 60 | 21 | 21 | 42
  61 - 70 | 27 | 24 | 51
  71 - 80 | 28 | 16 | 44
  81 + | 4 | 6 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 56 | 109
  Male | 53 | 43 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 92 | 84 | 176
  Unknown or Not Reported | 7 | 11 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Black or African American | 21 | 20 | 41
  White | 77 | 68 | 145
  Unknown or not reported | 6 | 10 | 16
Respiratory Support [Count of Participants; unit: Participants]
  On mechanical ventilation | 81 | 75 | 156
  On NIV | 5 | 3 | 8
  On HFNC | 20 | 21 | 41
  Missing | 0 | 0 | 0
CoVID Infected [Count of Participants; unit: Participants]
  Yes | 9 | 17 | 26
  No | 97 | 82 | 179

OUTCOME MEASURES:

1. Primary Outcome: Respiratory-support-free Days in Immunocompetent Patients With Sepsis-associated Acute Respiratory Failure
Description: To evaluate whether administration of ganciclovir increases respiratory-support-free days in immunocompetent patients with sepsis-associated acute respiratory failure. The outcome is the number of days the participant is not on respiratory support in the first 28 study days. This outcome uses the last-off approach to calculate the number of respiratory support days. The number of support days after calculated from the last day the participant was on respiratory support.
Time Frame: up to 28 days
Population: All participants enrolled, eligible, and evaluable (not replaced) and included in this primary analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 105 | 96
days | 12.1 (11.1) | 14.6 (10.5)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; The null hypothesis is that there is no significant difference in the number of respiratory support free days between the active drug arm and the placebo drug arm based on the student's t-test; Test type: Superiority; p = 0.098, t-test, 2 sided

2. Secondary Outcome: To Evaluate Whether Administration of Ganciclovir Increases Ventilator-free Days in Immunocompetent Patients With Sepsis-associated Acute Respiratory Failure.
Description: During the first 28 study days, the number of days the participants are not on mechanical ventilation using the last off approach is compared between the two treatment arms.
Time Frame: up to 28 study days
Population: Only the participants on mechanical ventilation at study entry are included. Participants on other types of respiratory support are excluded from this endpoint analysis.
Measure: Mean (Standard Deviation); unit: days not on mechanical ventilation
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 80 | 73
days not on mechanical ventilation | 11.7 (11.1) | 15.3 (10.6)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Superiority; p = 0.040, t-test, 2 sided

3. Secondary Outcome: To Evaluate Whether Administration of Ganciclovir Increases Total Respiratory-support-free Days (All RSFDS, Instead of Last-off Approach) in Immunocompetent Patients With Sepsis- Associated Acute Respiratory Failure
Description: During the first 28 study days, the number of days the participants are not on any respiratory-support is compared between the two treatment arms. Instead of using last-off approach, we will count all the days during 28 days period.
Time Frame: up to 28 days
Population: All participants enrolled, eligible, and evaluable (not replaced) and included in this primary analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 105 | 96
days | 12.9 (11.1) | 15.2 (10.2)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.130, t-test, 2 sided

4. Secondary Outcome: To Evaluate Whether Mortality and Time to Death in the 28 Days is Different Among Ganciclovir Recipients Relative to Placebo Recipients, Respectively.
Description: This is a time to event outcome with death as the event and censoring at the time of study termination if the participant is alive at 28 days. The hazard ratio and Cox proportional hazards models are used for this endpoint.
Time Frame: at study day 28
Population: Includes all participant enrolled, eligible, and evaluable (not replaced).
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 106 | 99
Participants | 34 | 13
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; The null hypothesis is that there is no difference between the two arms. The placebo arm is the comparison group; Test type: Superiority; p = 0.003, Regression, Cox; Hazard Ratio (HR) = 2.65, 95% CI 2-sided [1.40 to 5.02] — The placebo arm is the comparison arm (denominator). The incidence rate uses the person-years at risk for each of the study arms

5. Secondary Outcome: To Evaluate Whether Mortality and Time to Death in the 180 Days is Different Among Ganciclovir Recipients Relative to Placebo Recipients, Respectively.
Description: This is a time to event outcome with death as the event and censoring at the time of study termination if the participant is alive at the end of the study (day 180).
Time Frame: at the final study visit (day 180)
Population: Includes all participant enrolled, eligible, and evaluable (not replaced).
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 106 | 99
Participants | 45 | 22
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; the null hypothesis is that there is no difference between the two arms. The placebo group is the comparator group; Test type: Superiority; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 2.21, 95% CI 2-sided [1.32 to 3.68] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: To Evaluate Whether Duration of Mechanical Ventilation Among Survivors in the First 28 Days is Different Among Ganciclovir Recipients Relative to Placebo Recipients.
Description: This endpoint summarizes the days of mechanical ventilation for those participants who survive the first 28 days of the study. Participants who die in the first 28 days are excluded.
Time Frame: up to 28 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days on mechanical ventilation
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 52 | 62
days on mechanical ventilation | 10.0 (8.7) | 10.4 (9.3)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Superiority; p = 0.83, t-test, 2 sided

7. Secondary Outcome: To Evaluate Whether Duration of Respiratory Support Among Survivors in the First 28 Days is Different Among Ganciclovir Recipients Relative to Placebo Recipients.
Description: This endpoint summarizes the days of all types of respiratory support for those participants who survive the first 28 days of the study. Participants who die in the first 28 days are excluded.
Time Frame: up to 28 days
Population: Participants who survive the first 28 days of this study are included.
Measure: Mean (Standard Deviation); unit: days on respiratory support
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 71 | 82
days on respiratory support | 10.1 (8.8) | 11.2 (9.3)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Superiority; p = 0.457, t-test, 2 sided

8. Secondary Outcome: To Evaluate Whether Oxygenation is Different Among Ganciclovir Recipients Relative to Placebo Recipients.
Description: The PaO2/FiO2 (P/F) ratio was used to define oxygenation. The P/F ratio was summarized over the first 7 days of the study. The lowest PaO2 value within each study day was reported and used in the oxygenation calculation. If the PaO2 value was not available, an estimate of PaO2 was calculated from the SpO2 lowest value.
Time Frame: up to 7 days
Measure: Mean (Standard Deviation); unit: PaO2/FiO2
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 106 | 99
PaO2/FiO2
  Oxygenation Day 1 | 155.4 (78.4) | 184.8 (132.9)
  Oxygenation Day 2 | 177.3 (78.3) | 186.8 (112.2)
  Oxygenation Day 3 | 178.9 (72.0) | 186.8 (106.5)
  Oxygenation Day 4 | 190.5 (87.8) | 189.4 (79.1)
  Oxygenation Day 5 | 184.6 (80.3) | 196.3 (80.5)
  Oxygenation Day 6 | 209.1 (80.8) | 199.1 (106.6)
  Oxygenation Day 7 | 193.5 (81.1) | 198.5 (88.2)

9. Secondary Outcome: To Evaluate Whether ICU-free Days in the First 28 Days Are Different Among Ganciclovir Recipients Relative to Placebo Recipients.
Description: During the first 28 study days, the number of days the participants are not in ICU using the last off approach is compared between the two treatment arms.
Time Frame: up to 28 days
Population: All participants enrolled, eligible, and evaluable (not replaced) and included in this primary analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 105 | 95
days | 10.9 (10.4) | 13.9 (9.7)
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; The null hypothesis is that there is no significant difference in the number of ICU free days between the active drug arm and the placebo drug arm based on the student's t-test; Test type: Superiority; p = 0.037, t-test, 2 sided

10. Secondary Outcome: To Evaluate Whether CMV DNA Detection in Plasma and Endotracheal Aspirate (ETA) by Day 28 is Different Among Ganciclovir Recipients Relative to Placebo Recipients.
Description: CMV DNA detection in plasma and endotracheal aspirate (ETA) by day 28 is defined as positive CMV PCR result from any ETA, plasma, or serum specimen collected through day 28. CMV reactivation by day 28 will be summarized with number of participants with CMV reactivation in two levels: as any detectable CMV DNA (any level) and as high-level reactivation (>1000 IU/mL) for CMV negative patients at baseline.
Time Frame: up to 28 days
Population: Participants who tested CMV negative at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 85 | 77
Participants
  Any CMV reactivation | 5 | 20
  > 1000 UI/mL | 1 | 0
Statistical Analysis 1: Comparison: IV Ganciclovir vs Placebo; Test type: Superiority; p < 0.001, Fine-Gray competing risks regression — This analysis evaluated any level of CMV reactivation; This analysis will include death as a competing risk if it occurs on the same day of the last negative CMV test date
Statistical Analysis 2: Comparison: IV Ganciclovir vs Placebo; Test type: Superiority; p = 0.3, Fine-Gray competing risks regression — This analysis evaluate CMV reactivation > 1000 UI/mL; This analysis will include death as a competing risk if it occurs on the same day of the last negative CMV test date

11. Secondary Outcome: To Assess the Number and Severity of Adverse Events and Serious Adverse Events in the First 28 Days in Both Groups.
Description: During the first 28 days, this endpoint summarizes the number of participants who experienced adverse events (AEs) of severity grade ≥3 and whether any serious adverse events (SAEs) occurred in each study arm.
Time Frame: up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | IV Ganciclovir | Placebo
Number analyzed (Participants) | 106 | 99
Participants
  Participants with at least one reportable AE of grade 3 or greater | 13 | 11
  Participants with at least one SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to study final visit (180 days)
Description: Because critically ill patients exhibit numerous expected abnormalities, this study used a modified definition of reportable adverse events. A reportable AE is any clinically important untoward medical occurrence that (1) differs from what is expected, or (2) is considered related to the study drug or procedures, regardless of expectedness. More detail can be found in Protocol section 11.1. Note, most deaths were not reportable AEs but all deaths are included in the All Cause Mortality results.
Arm/Group | IV Ganciclovir | Placebo
All-Cause Mortality (participants affected / at risk) | 45/106 | 22/99
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/99
Other Adverse Events (participants affected / at risk) | 22/106 | 18/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Ganciclovir (N=106) | Placebo (N=99)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Acute cardiac event (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Subacute inflammatory demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Protocol (2025-07-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT04706507/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2025-10-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT04706507/SAP_002.pdf
  • Informed Consent Form (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/07/NCT04706507/ICF_000.pdf